CLINICAL TRIAL: NCT02047461
Title: A Phase 2, Multicenter, Multinational, Open-Label, Dose-Escalation Study to Evaluate the Safety and Efficacy of ORGN001 (Formerly ALXN1101) in Pediatric Patients With Molybdenum Cofactor Deficiency (MoCD) Type A Currently Treated With Recombinant Escherichia Coli-derived Cyclic Pyranopterin Monophosphate (rcPMP)
Brief Title: Safety & Efficacy Study of ORGN001 (Formerly ALXN1101) in Pediatric Patients With MoCD Type A Currently Treated With rcPMP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Origin Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1101-MCD-201; 2013-002701-56 (EudraCT Number)
Record Dates: First submitted 2014-01-09; First posted 2014-01-28 (Estimated); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Molybdenum Cofactor Deficiency, Type A
Keywords: Molybdenum cofactor deficiency (MoCD); molybdenum cofactor (MoCo) biosynthesis; sulfite oxidase (SO); xanthine dehydrogenase; aldehyde oxidase; S sulfocysteine (SSC)
MeSH Terms: conditions — Molybdenum Cofactor Deficiency, Complementation Group A; Molybdenum cofactor deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ORGN001 (formerly ALXN1101) (Experimental): daily IV infusions
  Interventions: Drug: ORGN001 (formerly ALXN1101)

INTERVENTIONS:
Drug: ORGN001 (formerly ALXN1101) — IV infusion

SUMMARY:
This study will include a screening period, a 6-month treatment period, followed by long-term extension period expected to last approximately 72 months.

DETAILED DESCRIPTION:
Patients will receive daily IV infusions of ORGN001 (formerly ALXN1101) starting on Day 1. After a prescribed period, dosing will increase monthly based on defined patient safety measures. After Month 6, patients will continue daily dosing at their last tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with a genetically confirmed diagnosis of MoCD Type A (MOCS1 mutation)
* Currently treated with rcPMP infusions

Exclusion Criteria:

- Current or planned treatment with another investigational drug or device, with the exception rcPMP treatment through Day -1.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States
- Monash Medical Centre, Melbourne, Australia
- Beatrix Children's Hospital, Groningen, Netherlands
- Unité des maladies métaboliques, Tunis, Tunisia
- United Kingdom (2):
  - Royal Hospital for Sick Children, Glasgow
  - Manchester University Hospitals NHS Foundation Trust, Manchester

REFERENCES:
- See also: FDA Drug Approval Package — https://www.accessdata.fda.gov/drugsatfda_docs/nda/2021/214018Orig1s000TOC.cfm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who were currently receiving rcPMP infusions were enrolled and transitioned to ORGN001.
Groups:
- Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001: Patients currently receiving rcPMP infusions at baseline are transitioned to ORGN001 (formerly ALXN1101), starting at their current rcPMP dose and escalating to a target cPMP dose of 0.9 mg/kg.
Period: Overall Study
Arm/Group | Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients currently receiving rcPMP infusions at Baseline and transitioned to ORGN001.
Groups:
- Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001: Patients currently receiving rcPMP infusions at baseline are transitioned to ORGN001 (formerly ALXN1101), starting at their current rcPMP dose and escalating to a target dose of cPMP 0.9 mg/kg per protocol
Arm/Group | Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 45.2 (22.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 2
  United States | 1
  United Kingdom | 3
  Australia | 1
  Tunisia | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of ORGN001 (Formerly ALXN1101)
Description: Treatment Emergent Serious Adverse Events
Time Frame: Baseline to Month 24 for all patients plus additional follow-up up to Month 90
Population: Full Analysis Set
Measure: Number; unit: events
Groups:
- Patient Currently Receiving rcPMP Infusions at Baseline: Patient currently receiving rcPMP infusions at Baseline and transitioned to ORGN001
Arm/Group | Patient Currently Receiving rcPMP Infusions at Baseline
Number analyzed (Participants) | 8
events
  Gastrointestinal disorders | 1
  General disorders and administration site conditions | 5
  Infections and infestations | 6
  Injury, poisoning and procedural complications | 2
  Metabolism and nutrition disorders | 2
  Musculoskeletal and connective tissue disorders | 1
  Nervous system disorders | 2
  Product issues | 1
  Respiratory, thoracic and mediastinal disorders | 2
  Skin and subcutaneous tissue disorders | 1
  Surgical and medical procedures | 1
  Vascular disorders | 2

2. Secondary Outcome: Pharmacokinetics (Actual Plasma Concentration) of ORGN001 (Formerly ALXN1101)
Description: ORGN001 levels by dose at pre-infusion and end of infusion (EOI) at scheduled timepoints
Time Frame: First 6 months at each dose level, where available
Population: Measurement is actual plasma concentration of ORGN001 at measured timepoints, starting at their current rcPMP dose. 6 patients started at a dose of 240 mcg/kg, 1 patient at 248 mcg/kg, and 1 patient at 280 mcg/kg. (EOI = End of Infusion). 1 patient is missing a pre-infusion dose measurement.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001: Patients currently receiving rcPMP infusions at baseline are transitioned to ORGN001 (formerly ALXN1101), starting at their current rcPMP dose and escalating to a target dose of 0.9 mg/kg
Arm/Group | Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001
Number analyzed (Participants) | 8
ng/mL
  Day 1 Pre-infusion (240 mcg/kg): number analyzed (Participants) | 6
  Day 1 Pre-infusion (240 mcg/kg) | 3.95 (9.68)
  Day 1 Pre-infusion (248 mcg/kg): number analyzed (Participants) | 1
  Day 1 Pre-infusion (248 mcg/kg) | 0 (NA) — There is only one patient with data and therefore there is no Standard Deviation.
  Day 1 EOI (240 mcg/kg): number analyzed (Participants) | 6
  Day 1 EOI (240 mcg/kg) | 669.00 (236.06)
  Day 1 EOI (248 mcg/kg): number analyzed (Participants) | 1
  Day 1 EOI (248 mcg/kg) | 36.00 (NA) — There is only one patient with data and therefore there is no Standard Deviation.
  Day 1 EOI (280 mcg/kg): number analyzed (Participants) | 1
  Day 1 EOI (280 mcg/kg) | 770.00 (NA) — There is only one patient with data and therefore there is no Standard Deviation.
  Day 7 EOI (240 mcg/kg): number analyzed (Participants) | 6
  Day 7 EOI (240 mcg/kg) | 699.50 (246.72)
  Day 7 EOI (248 mcg/kg): number analyzed (Participants) | 1
  Day 7 EOI (248 mcg/kg) | 694.00 (NA) — There is only one patient with data and therefore there is no Standard Deviation.
  Day 60 EOI (480 mcg/kg): number analyzed (Participants) | 5
  Day 60 EOI (480 mcg/kg) | 880.84 (558.56)
  Day 90 EOI (240 mcg/kg): number analyzed (Participants) | 1
  Day 90 EOI (240 mcg/kg) | 1230.00 (NA) — There is only one patient with data and therefore there is no Standard Deviation.
  Day 90 EOI (480 mcg/kg): number analyzed (Participants) | 1
  Day 90 EOI (480 mcg/kg) | 762.00 (NA) — There is only one patient with data and therefore there is no Standard Deviation.
  Day 90 EOI (720 mcg/kg): number analyzed (Participants) | 6
  Day 90 EOI (720 mcg/kg) | 1888.33 (271.10)
  Day 120 EOI (480 mcg/kg): number analyzed (Participants) | 1
  Day 120 EOI (480 mcg/kg) | 2810.00 (NA) — There is only one patient with data and therefore there is no Standard Deviation.
  Day 120 EOI (720 mcg/kg): number analyzed (Participants) | 1
  Day 120 EOI (720 mcg/kg) | 671.00 (NA) — There is only one patient with data and therefore there is no Standard Deviation.
  Day 120 EOI (960 mcg/kg): number analyzed (Participants) | 6
  Day 120 EOI (960 mcg/kg) | 4213.33 (4520.31)
  Day 150 EOI (720 mcg/kg): number analyzed (Participants) | 1
  Day 150 EOI (720 mcg/kg) | 3810.00 (NA) — There is only one patient with data and therefore there is no Standard Deviation.
  Day 150 EOI (960 mcg/kg): number analyzed (Participants) | 3
  Day 150 EOI (960 mcg/kg) | 2045.67 (1009.84)
  Day 150 EOI (1200 mcg/kg): number analyzed (Participants) | 3
  Day 150 EOI (1200 mcg/kg) | 3173.33 (656.53)

3. Secondary Outcome: S-sulfocysteine (Umol/L) Normalized to Urine Creatinine (mmol/L) - Change From Baseline Over Time
Description: Analyses were performed on urine SSC, a biomarker of the MoCD pathway. Levels of SSC measured in urine were normalized to urine creatinine levels. The observed value, change, and percent change in urine and blood SSC levels from baseline were summarized by visit over time.
Time Frame: Baseline to Month 24 for all patients plus additional follow-up to Month 90
Population: Not all patients had samples taken at each expected timepoint.
Measure: Mean (Standard Deviation); unit: umol/mmol
Arm/Group | Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001
Number analyzed (Participants) | 8
umol/mmol
  Baseline | 21.1 (12.89)
  Day 4 Change from Baseline | -1.7 (12.70)
  Day 7 Change from Baseline | -7.8 (9.70)
  Day 14 Change from Baseline | -2.2 (14.51)
  Day 28 Change of Baseline: number analyzed (Participants) | 7
  Day 28 Change of Baseline | 2.8 (14.17)
  Day 57 Change from Baseline: number analyzed (Participants) | 7
  Day 57 Change from Baseline | -3.0 (10.29)
  Day 127 Change from Baseline | -12.2 (14.77)
  Month 6 Change from Baseline | -13.6 (11.77)
  Month 12 Change from Baseline | -8.6 (20.15)
  Month 24 Change from Baseline | -14.3 (14.73)
  Month 36 Change from Baseline: number analyzed (Participants) | 5
  Month 36 Change from Baseline | -13.2 (18.40)
  Month 48 Change from Baseline: number analyzed (Participants) | 5
  Month 48 Change from Baseline | -6.7 (6.65)
  Month 60 Change from Baseline: number analyzed (Participants) | 4
  Month 60 Change from Baseline | -17.9 (14.59)
  Month 90 Change from Baseline: number analyzed (Participants) | 2
  Month 90 Change from Baseline | 1.7 (10.25)

4. Secondary Outcome: Effect of ORGN001 (Formerly ALXN1101) on Neurologic Function Including Motor Examination
Description: Change from baseline on repeated Neurologic examinations such as muscle strength and tone, as well as sensory and reflex exam.
Time Frame: Baseline to Month 24 for all patients plus additional follow-up until Month 30
Population: All patients entering the study had complete examinations throughout the study to identify Normal vs Abnormal Neurologic Function on the parameters presented. Date shown here are from Baseline and final examination where all 8 patients have data.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001
Number analyzed (Participants) | 8
Participants
  Quality of Spontaneous Movement at Baseline: Normal | 3
  Quality of Spontaneous Movement at Baseline: Abnormal | 5
  Quality of Spontaneous Movement at Month 30: Normal | 4
  Quality of Spontaneous Movement at Month 30: Abnormal | 4
  Dystonic at Baseline: Normal | 4
  Dystonic at Baseline: Abnormal | 4
  Dystonic at Month 30: Normal | 4
  Dystonic at Month 30: Abnormal | 4
  Opistonic at Baseline: Normal | 7
  Opistonic at Baseline: Abnormal | 1
  Opistonic at Month 30: Normal | 6
  Opistonic at Month 30: Abnormal | 2
  Truncal Tone at Baseline: number analyzed (Participants) | 7
  Truncal Tone at Baseline: Normal | 2
  Truncal Tone at Baseline: Abnormal | 5
  Truncal Tone at Month 30: Normal | 2
  Truncal Tone at Month 30: Abnormal | 6
  Appendicular Tone at Baseline: Normal | 2
  Appendicular Tone at Baseline: Abnormal | 6
  Appendicular Tone at Month 30: Normal | 1
  Appendicular Tone at Month 30: Abnormal | 7
  Deep Tendon reflexes at Baseline: Normal | 4
  Deep Tendon reflexes at Baseline: Abnormal | 4
  Deep Tendon reflexes at Month 30: Normal | 3
  Deep Tendon reflexes at Month 30: Abnormal | 5
  Primitive reflexes at Baseline: number analyzed (Participants) | 6
  Primitive reflexes at Baseline: Normal | 5
  Primitive reflexes at Baseline: Abnormal | 1
  Primitive reflexes at Month 30: number analyzed (Participants) | 7
  Primitive reflexes at Month 30: Normal | 6
  Primitive reflexes at Month 30: Abnormal | 1
  Clonus presence at Baseline: Normal | 7
  Clonus presence at Baseline: Abnormal | 1
  Clonus presence at Month 30: Normal | 6
  Clonus presence at Month 30: Abnormal | 2
  Ambulation at Baseline: Normal | 4
  Ambulation at Baseline: Abnormal | 4
  Ambulation at Month 30: Normal | 4
  Ambulation at Month 30: Abnormal | 4

5. Secondary Outcome: Long-term Safety of ORGN001 (Formerly ALXN1101)
Description: Change from baseline in Seizure frequency
Time Frame: Baseline to Month 24 for all patients plus additional follow up until Month 72
Population: Number of patients with Seizures in observation period
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001
Number analyzed (Participants) | 8
Participants
  Screening: number analyzed (Participants) | 7
  Screening | 3
  Baseline to Month 6: number analyzed (Participants) | 7
  Baseline to Month 6 | 4
  Month 6 to Month 12 | 3
  Month 12 to Month 24 | 3
  Month 24 to Month 36 | 3
  Month 36 to Month 48: number analyzed (Participants) | 7
  Month 36 to Month 48 | 3
  Month 48 to Month 60: number analyzed (Participants) | 7
  Month 48 to Month 60 | 3
  Month 60 to Month 72: number analyzed (Participants) | 7
  Month 60 to Month 72 | 3

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 1 with ORGN001 treatment until Month 24 for all patients; additional data included for patients treated up to Month 90
Description: All-cause Mortality is zero in this study because there were no deaths that occurred.
  All SAE data is included
Arm/Group | Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 8/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001 (N=8)
Complication associated with device (General disorders) | 4
Pyrexia (General disorders) | 2
Catheter site infections (Infections and infestations) | 2
Device related infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Vascular device infection (Infections and infestations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Currently Receiving rcPMP Infusions at Baseline and Transitioned to ORGN001 (N=8)
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1
Chalazion (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Eye swelling (Eye disorders) | 2
Strabismus (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Barrett's oesophagus (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Noninfective gingivitis (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1
Teething (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Catheter site discharge (General disorders) | 2
Catheter site discoloration (General disorders) | 1
Catheter site extravasation (General disorders) | 2
Catheter site haemorrhage (General disorders) | 1
Catheter site irritation (General disorders) | 1
Catheter site oedema (General disorders) | 1
Catheter site pain (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Complication associated with device (General disorders) | 6
Gait disturbance (General disorders) | 1
Medical device site discomfort (General disorders) | 1
Medical device site reaction (General disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 7
Swelling (General disorders) | 1
Swelling face (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Blister infected (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
Bullous impetigo (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 2
Catheter site abscess (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Ear infection (Infections and infestations) | 2
Ear infection viral (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 2
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 4
Lower respiratory tract infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 3
Otitis media acute (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 4
Pneumonia influenzal (Infections and infestations) | 1
Pustule (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Urinary tract infection bacterial (Infections and infestations) | 1
Varicella (Infections and infestations) | 2
Vascular device infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 5
Viral tonsillitis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 2
Muscle injury (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Scar (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Blood iron decreased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Cardiac murmur (Investigations) | 1
Culture urine positive (Investigations) | 1
Heart rate increased (Investigations) | 1
Procalcitonin increased (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 2
Growth retardation (Musculoskeletal and connective tissue disorders) | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral atrophy (Nervous system disorders) | 1
Dystonia (Nervous system disorders) | 1
Dystonia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Hypertonia (Nervous system disorders) | 1
Muscle spasticity (Nervous system disorders) | 1
Opisthotonos (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Tonic convulsion (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Device dislocation (Product Issues) | 3
Device leakage (Product Issues) | 2
Device occlusion (Product Issues) | 1
Agitation (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Acute respiratory failure (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
This was an open label study with no comparator arm. Limited statistical analysis were performed. Most data was summarized over time by individual patient, making reportable results in tabular format truncated. Refer to FDA approval package for more information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/Investigator shall have the right to publish or present the results of Institution's and Investigator's activities including that Study Data which was obtained or derived at Institution. Institution/ Investigator agree to submit any proposed publication/presentation to Sponsor for review at least 60 days prior to submitting any such proposed publication. Within 30 days of its receipt, Sponsor shall advise if any changes are needed to protect confidentiality.

DOCUMENTS (2):
  • Study Protocol (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT02047461/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT02047461/SAP_001.pdf